CLINICAL TRIAL: NCT00497705
Title: Genes Causing Congenital Ebstein's Anomaly
Brief Title: Genes Causing Ebstein's Anomaly
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070186; 07-H-0186
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-07-07

CONDITIONS: Heart Septal Defects, Ventricle; Heart Defects, Congenital; Double Outlet Right Ventricle; Truncus Arteriosus, Persistent
Keywords: Ebsteins Anomaly; Heart Septal Defects, Ventricle; Heart Defects, Congenital; Double Outlet Right Ventricle; Truncus Arteriosus Persistant; Ebstein's Anomaly; Congenital Heart Disease; Heart Defects
MeSH Terms: conditions — Heart Septal Defects; Heart Defects, Congenital; Double Outlet Right Ventricle; Truncus Arteriosus, Persistent; Ebstein Anomaly

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will investigate Ebstein's anomaly, a congenital abnormality of the tricuspid valve of the heart and try to identify the genetic origins of the disease.

Adults and children 2 years of age and older with Ebstein's anomaly and healthy volunteers may be eligible for this study. Participants undergo the following procedures:

* Blood tests: Three tube of blood will be collected, with the total amount limited to about half a teaspon for each two pounds of body weight.
* Saliva sample collection: A small amount of saliva is collected by spitting into a sterile container.
* Oral (cheek) swab: Cells are collected from the mouth using a soft brush to swab the inside lining of the cheek.
* Electrocardiogram: The electrical activity of the heart is recorded using electrodes placed on the chest.
* Echocardiogram: Heart function is assessed using ultrasound.

DETAILED DESCRIPTION:
The goal of this study is to elucidate the genetic basis for the congenital heart disease (CHD) known as Ebstein's anomaly. These studies complement ongoing research studies using mouse models to recover mutations causing structural heart defects associated with human CHD. By elucidating the underlying genetic causes for Ebstien's anomaly, it may be possible to improve risk assessments as well as facilitate the development of new strategies for prevention and disease management. These studies are important for early diagnosis and the management of complications associated with surviving adults with Ebstein's anomaly, some of whom have undergone surgical correction and others that are unoperated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients who have diagnosed Ebstein's anomaly or tricuspid valve disease in Belarus or Ukraine and their parents will be asked to participate in this study regardless of sex, age, or race. In addition, sex and age matched neighborhood children and their parents will be recruited as controls. There is no known ethnic or racial predilection for Ebstein's anomaly or tricuspid valve disease.

EXCLUSION CRITERIA:

There are no exclusion criteria. This may allow us to discover previously unknown relationships between Ebstein's anomaly and other diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-07-03; Primary Completion 2009-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Republican Scientific and Clinical Cardiology Center, Republic of Belarus, Belarus
- Amosov Institute of Cardiovascular Surgery, Kyiv, Ukraine

REFERENCES:
- [Background] Abu-Issa R, Waldo K, Kirby ML. Heart fields: one, two or more? Dev Biol. 2004 Aug 15;272(2):281-5. doi: 10.1016/j.ydbio.2004.05.016. No abstract available. PMID 15282148
- [Background] Attenhofer Jost CH, Connolly HM, Dearani JA, Edwards WD, Danielson GK. Ebstein's anomaly. Circulation. 2007 Jan 16;115(2):277-85. doi: 10.1161/CIRCULATIONAHA.106.619338. No abstract available. PMID 17228014
- [Background] Basson CT, Bachinsky DR, Lin RC, Levi T, Elkins JA, Soults J, Grayzel D, Kroumpouzou E, Traill TA, Leblanc-Straceski J, Renault B, Kucherlapati R, Seidman JG, Seidman CE. Mutations in human TBX5 [corrected] cause limb and cardiac malformation in Holt-Oram syndrome. Nat Genet. 1997 Jan;15(1):30-5. doi: 10.1038/ng0197-30. PMID 8988165